CLINICAL TRIAL: NCT05532657
Title: Long-term Effects of Hearing Intervention on Brain Health in the Aging and Cognitive Health Evaluation in Elders Randomized Study
Brief Title: ACHIEVE Brain Health Follow-Up Study
Acronym: ACHIEVE-BHFU
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of North Carolina (Other); University of South Florida (Other); University of Minnesota (Other); University of Mississippi Medical Center (Other); Wake Forest University (Other); Mayo Clinic (Other); National Institute on Aging (NIA) (NIH); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00319430; R01AG076518 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Aging; Cognitive Decline; Mild Cognitive Impairment; Dementia; Hearing Loss
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Hearing Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing intervention (HI) group (Active Comparator): Participants in this group were randomized to the hearing intervention (HI) group at ACHIEVE trial baseline and received a best practices hearing rehabilitation treatment program, consisting of fitting with hearing aids and other hearing assistive technologies along with comprehensive, individualized hearing rehabilitation sessions with a study audiologist spaced over the 2-3 months post-fitting designed to provide all the active components of the intervention. Participants also received semi-annual booster sessions with the study audiologist. These participants will continue to receive hearing healthcare from the study audiologist and complete semi-annual sessions for 3 additional years.
  Interventions: Other: Hearing intervention
- Successful aging/Delayed hearing intervention (SA/DHI) group (Active Comparator): Participants in this active control group were randomized to the successful aging (SA) group at ACHIEVE trial baseline and received a successful aging health education program, following the protocol and materials developed for the 10 Keys to Healthy Aging program. The program involved individualized sessions with a study health educator to control for staff-participant time and attention between the two groups. Upon completion of the ACHIEVE trial, these participants are offered the best practices hearing rehabilitative treatment program with comprehensive, individualized sessions post-fitting and will receive semi-annual booster sessions with the study audiologist for 3 years.
  Interventions: Other: Successful aging/delayed hearing intervention

INTERVENTIONS:
Other: Hearing intervention — The hearing intervention is best practices hearing rehabilitation treatment program, consisting of fitting with hearing aids and other hearing assistive technologies along with comprehensive, individualized hearing rehabilitation sessions with a study audiologist spaced over the 2-3 months post-fitting designed to provide all the active components of the intervention. Participants also received semi-annual booster sessions with the study audiologist for 3 years and will continue to receive hearing healthcare from the study audiologist and complete semi-annual sessions for 3 additional years.
  Arms: Hearing intervention (HI) group
Other: Successful aging/delayed hearing intervention — The successful aging health education program follows the protocol and materials developed for the 10 Keys to Healthy Aging program. The program involved individualized sessions with a study health educator, with initial sessions spaced over the 2-3 months post-randomization and semi-annual sessions for 3 years. Upon completion of the ACHIEVE trial, these participants are offered the best practices hearing rehabilitative treatment program with comprehensive, individualized sessions post-fitting and will receive semi-annual booster sessions with the study audiologist for 3 years.
  Arms: Successful aging/Delayed hearing intervention (SA/DHI) group

SUMMARY:
The ACHIEVE Brain Health Follow-Up Study is a 3-year follow-up to the Aging and Cognitive Health Evaluation in Elders (ACHIEVE) randomized study to determine the long-term effect of hearing intervention vs. successful aging/delayed hearing intervention on rates of cognitive decline and incident mild cognitive impairment or dementia.

DETAILED DESCRIPTION:
ORIGINAL ACHIEVE TRIAL:

The Aging and Cognitive Health Evaluation in Elders (ACHIEVE) study is an National Institute on Aging (NIA)-sponsored Phase III randomized controlled trial (R01AG055426; Multiple Principal Investigators: Lin/Coresh) investigating whether hearing loss treatment versus an aging education control intervention reduces cognitive decline over a 3-year follow-up period. From 2018 to 2019, the investigators recruited 977 adults aged 70-84 years with untreated mild-to-moderate hearing loss who were randomized 1:1 at baseline to receive hearing intervention (HI; best practices hearing services and technologies) versus a successful aging (SA) education control intervention (i.e., one-on-one sessions with a health educator covering topics important for healthy aging). Participants are followed semi-annually at the ACHIEVE field sites (Washington County, Maryland; Jackson, Mississippi; Minneapolis, Minnesota; Forsyth County; North Carolina) with final Year 3 study visits for ACHIEVE participants scheduled from 2021-2022. After the participants Year 3 visit, all participants randomized to the SA education control group will also be offered the hearing intervention. Final Year 3 results from this original trial will indicate whether hearing intervention (versus a successful aging control intervention) reduces cognitive decline over a 3-year interval after randomization.

ACHIEVE BRAIN HEALTH FOLLOW-up STUDY:

The current study will continue following the ACHIEVE cohort for an additional 3 years after the participants Year 3 visit (i.e., total of 6 years) to determine the long-term effects of hearing intervention (i.e., participants randomized to HI at ACHIEVE baseline) versus successful aging/delayed HI control (i.e., participants randomized to SA at ACHIEVE baseline and offered HI after the participants ACHIEVE Year 3 visit) on cognitive, dementia, and brain outcomes. Given that cognitive impairment typically reflects the slow accumulation of pathologic changes, the benefits of hearing intervention in slowing this decline may not be fully appreciable within just 3 years. Therefore, this 6-year follow-up of the cohort will allow the investigators to fully evaluate the longer, cumulative impact of hearing loss treatment on older adults. Such findings will complement the main trial results in 2023 and directly inform clinical and policy decisions around the potential use of hearing interventions to reduce the risk of cognitive decline and Alzheimer's disease and related dementias (ADRD).

ELIGIBILITY:
To be eligible for ACHIEVE-BHFU, participants must meet the following criteria:

* Eligible for and participated in the ACHIEVE trial (see original criteria below)
* Agree to participate and are able and willing to comply with study procedures for three years in the follow-up study

Original ACHIEVE Inclusion Criteria (during 2018-2019 enrollment):

* Age 70-84 years
* Community dwelling, fluent English speaker
* Availability of participant in area for study duration
* Adult-onset hearing impairment, defined as four-frequency pure tone average (PTA, 0.5-4 kilohertz (kHz), better ear) ≥ 30 decibels hearing level (dB HL) & ≤ 70 dB HL
* Speech recognition scores in quiet ≥ 60% in better ear
* Mini-Mental State Exam (MMSE) score ≥ 23 for high school degree or less; ≥ 25 for some college or more

Original ACHIEVE Exclusion Criteria:

* Reported disability in ≥ 2 activities of daily living (ADLs)
* Vision impairment (worse than 20/63 on the Minnesota Near Vision Card)
* Self-reported use of a hearing aid in the past 1 year
* Medical contraindication to use of hearing aids (e.g., draining ear)
* Unwilling to wear hearing aids on a daily basis
* Conductive hearing impairment with air-bone gap > 15 dB (decibels) in two or more contiguous frequencies in both ears

Min Age: 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 629 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in global cognition | ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years)
  Change from original ACHIEVE trial baseline to ACHIEVE-BHFU final visit in global cognition, as assessed using a factor score derived from completion of a neurocognitive testing battery. The ACHIEVE and ACHIEVE Brain Health studies administer a neurocognitive testing battery annually, which includes the following cognitive tests: Delayed Word Recall, Incidental Learning, Logical Memory I and II, Word Fluency, Animal Naming, Boston Naming, Trail Making Test A and B, Digit Span Backwards, and Digit Symbol Substitution. Factor analytic methods use all items from all tests in the battery to generate a single global cognition score.
Mild cognitive impairment (MCI) / dementia | 6 years
  Time until composite outcome of adjudicated diagnosis of mild cognitive impairment (MCI) or dementia over the course of follow-up from original ACHIEVE trial baseline until ACHIEVE-BHFU final visit.

SECONDARY OUTCOMES:
Change in cognition memory domain | ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years)
  Change from original ACHIEVE trial baseline to ACHIEVE-BHFU final visit in the cognition memory domain, as assessed using a memory domain factor score derived from completion of a neurocognitive testing battery. The cognitive tests for the memory domain include Delayed Word Recall, Incidental Learning, and Logical Memory I and II. These tests have an underlying commonality, or factor, that is unable to be directly measured, and factor analytic methods use items from the tests noted to generate a single overall memory score.
Change in cognition executive function domain | ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years)
  Change from original ACHIEVE trial baseline to ACHIEVE-BHFU final visit in the cognition executive function domain, as assessed using an executive function domain factor score derived from completion of a neurocognitive testing battery. The cognitive tests for the executive function domain include Trail Making Test A and B and Digit Symbol Substitution. These tests have an underlying commonality, or factor, that is unable to be directly measured, and factor analytic methods use items from the tests noted to generate a single overall executive function score.
Change in cognition language domain | ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years)
  Change from original ACHIEVE trial baseline to ACHIEVE-BHFU final visit in the cognition language domain, as assessed using a language domain factor score derived from completion of a neurocognitive testing battery. The cognitive tests for the language domain include Word Fluency, Animal Naming, and Boston Naming. These tests have an underlying commonality, or factor, that is unable to be directly measured, and factor analytic use items from the tests noted to generate a single overall language score.
Change in regional brain volumes | If in ACHIEVE-MRI: ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years); if not in ACHIEVE-MRI: ACHIEVE-BHFU Baseline, ACHIEVE-BHFU Year 3 (~2.5 years)
  Change in volume (cm^3) of each MRI-defined brain region of interest from ACHIEVE trial baseline to ACHIEVE-BHFU final visit if the participant previously participated in the ACHIEVE-MRI ancillary study, or from ACHIEVE-BHFU baseline visit to ACHIEVE-BHFU final visit if the participant was not previously enrolled in the ACHIEVE-MRI ancillary study.
Change in white matter tract integrity | If in ACHIEVE-MRI: ACHIEVE Baseline, ACHIEVE-BHFU Year 3 (~6 years); if not in ACHIEVE-MRI: ACHIEVE-BHFU Baseline, ACHIEVE-BHFU Year 3 (~2.5 years)
  Change in MRI fractional anisotropy and mean diffusivity in white matter tracts from ACHIEVE trial baseline to ACHIEVE-BHFU final visit if the participant previously participated in the ACHIEVE-MRI ancillary study, or from ACHIEVE-BHFU baseline visit to ACHIEVE-BHFU final visit if the participant was not previously enrolled in the ACHIEVE-MRI ancillary study.

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Lin, MD, PhD, Principal Investigator — Johns Hopkins University; Josef Coresh, MD, PhD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Johns Hopkins Comstock Center for Public Health Research and Prevention, Hagerstown, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The ACHIEVE Data Coordinating Center, in coordination with the Steering Committee and NIH, will prepare a public access data release that complies with prevailing NIH and HIPAA guidelines in place when the study has been completed. Any participant identifying information will be removed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share data 1 year following publication of the main results paper for the trial, unless NIH policy dictates that data be shared sooner.
Access Criteria: To be determined

REFERENCES:
- [Background] Gross AL, Power MC, Albert MS, Deal JA, Gottesman RF, Griswold M, Wruck LM, Mosley TH Jr, Coresh J, Sharrett AR, Bandeen-Roche K. Application of Latent Variable Methods to the Study of Cognitive Decline When Tests Change over Time. Epidemiology. 2015 Nov;26(6):878-87. doi: 10.1097/EDE.0000000000000379. PMID 26414855